CLINICAL TRIAL: NCT00456287
Title: Platelet Activation and Circadian Rhythms of Clotting-Fibrinolysis Factors in Patients With Sleep Apnea Syndrome. Implications in the Precipitation of Cardiovascular Events
Brief Title: Platelet Activation and Circadian Rhythms of Clotting-Fibrinolysis Factors in Patients With Sleep Apnea Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Fundacion Caubet-Cimera Islas Baleares (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-109
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Sleep Apnea; Cardiovascular Diseases
Keywords: Sleep Apnea; Clotting- fibrinolysis patterns; Platelet function markers; Endothelial dysfunction
MeSH Terms: conditions — Sleep Apnea Syndromes; Cardiovascular Diseases | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP (Continuous Positive Airway Pressure)

SUMMARY:
The objective of the study is to define and compare clotting- fibrinolysis patterns, platelet function markers and endothelial dysfunction in patients with SAHS before and after treatment and normal controls age and weight matched.

DETAILED DESCRIPTION:
The hypothesis of the study is the following: Patients with sleep apnea-hypopnea syndrome have higher risk of cardiovascular mortality during the night.

Respiratory alterations (hypoxia, hypoxia- reoxygenation) that these patients suffer during the sleep may induce modifications in platelet function, clotting-fibrinolysis factors and endothelial function, that may accelerate cardiovascular events during the night

DESIGN: Prospective and controlled study

METHODS: 20 SAHS patients and 20 controls will be studied. The study includes:

a) medical history; b) anthropometric variables (weight, height, body mass index, waist-hip ratio); c) sleepiness tested by Epworth scale; d) conventional polysomnography (PSG); e) testing every 4 hours for a 24 hours period: clotting-fibrinolysis factors (factor V, VII, VIII; C and S protein, plasminogen tissular activator (t-PA) and inhibitor of plasminogen activator (PAI-1); platelet activation markers (CD62, CD63 and GPIIb/IIIa) and endothelial dysfunction markers (endothelins, nitrites/nitrates and asymmetrical dimethyl-arginine); f) basic biochemical profile and hemogram. Patients will be revaluated after 6 months of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-Hypopnea Index > 15

Exclusion Criteria:

* Presence of any chronic disease
* Presence of cardiovascular disease
* Refusal to sign informed consent
* Drug addiction and/or alcoholism
* Any medication two weeks before

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-02

PRIMARY OUTCOMES:
To define and compare clotting- fibrinolysis patterns, platelet function markers and endothelial dysfunction

SECONDARY OUTCOMES:
CPAP (Continuous Positive Airway Pressure) effect on studied variables

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Barceló, MD, Principal Investigator — Hospital Universitario Son Dureta
Locations (1):
- Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands, Spain